CLINICAL TRIAL: NCT01217931
Title: Sequential Two-agent Assessment in Renal Cell Carcinoma Therapy: The START Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0085; NCI-2011-00256 (Registry Identifier: NCI CTRP-Clinical Trials Registry)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Kidney Cancer
Keywords: Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Clear cell component; RCC; Bevacizumab; Everolimus; Pazopanib; GW786034; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Afinitor; RAD001
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — pazopanib; Bevacizumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): Pazopanib + possible Bevacizumab
  Interventions: Drug: Pazopanib; Drug: Bevacizumab
- Group 2 (Experimental): Pazopanib + possible Everolimus
  Interventions: Drug: Pazopanib; Drug: Everolimus
- Group 3 (Experimental): Everolimus + possible Bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Everolimus
- Group 4 (Experimental): Everolimus + possible Pazopanib
  Interventions: Drug: Pazopanib; Drug: Everolimus
- Group 5 (Experimental): Bevacizumab + possible Pazopanib
  Interventions: Drug: Bevacizumab
- Group 6 (Experimental): Bevacizumab + possible Everolimus
  Interventions: Drug: Bevacizumab; Drug: Everolimus

INTERVENTIONS:
Drug: Pazopanib — 800 mg by mouth once daily for 28 days. A cycle consists of 4 weeks.
  Other Names: GW786034
  Arms: Group 1; Group 2; Group 4
Drug: Bevacizumab — 10 mg/kg by vein every two weeks. A cycle consists of 4 weeks.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
  Arms: Group 1; Group 3; Group 5; Group 6
Drug: Everolimus — 10 mg by mouth once daily. A cycle consists of 4 weeks.
  Other Names: Afinitor; RAD001
  Arms: Group 2; Group 3; Group 4; Group 6

SUMMARY:
The goal of this clinical research study is to compare 6 different 2-drug "sequences" of everolimus, bevacizumab, or pazopanib to learn how they may affect metastatic kidney cancer. For the 2-drug sequence, participants will receive 1 of these drugs and may start taking another of these drugs after that. Researchers will also study the safety of these 2-drug sequences.

DETAILED DESCRIPTION:
The Study Drugs:

Everolimus is designed to block the growth of cancer cells, which may cause cancer cells to die.

Bevacizumab is designed to block the growth of blood vessels that supply nutrients necessary for tumor growth. This may prevent or slow down the growth of cancer cells.

Pazopanib is designed to block a protein that may cause uncontrolled tumor growth. Blocking this protein may prevent cancer from growing and spreading.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to 1 of 6 groups. There is an equal chance of being assigned to each group.

* Group 1 will receive pazopanib, possibly followed by bevacizumab.
* Group 2 will receive pazopanib, possibly followed by everolimus.
* Group 3 will receive everolimus, possibly followed by bevacizumab.
* Group 4 will receive everolimus, possibly followed by pazopanib.
* Group 5 will receive bevacizumab, possibly followed by pazopanib.
* Group 6 will receive bevacizumab, possibly followed by everolimus.

If the disease gets worse while you receive your first assigned drug, you will stop taking the drug. Then if you are not having side effects, you will start taking your second assigned drug 2-4 weeks later.

Everolimus is taken by mouth 1 time per day (at about the same time each day).

Bevacizumab is given by vein over 30-90 minutes, 1 time every 2 weeks.

Pazopanib is taken by mouth 1 time per day (at about the same time each day on an empty stomach).

You may be able to receive the bevacizumab doses at your local doctor's office. Ask your study doctor about this.

Study Visits:

Every week during Weeks 1-4, your blood pressure will be checked (either at home, at the clinic, or by your local doctor) if you are taking pazopanib or bevacizumab. If you are checking your own blood pressure at home, you should keep a log to write down your blood pressure. Bring the log to your next clinic visit.

Every 2 weeks, urine will be collected for routine tests if you are receiving bevacizumab.

Every 4 weeks:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking.
* You will be asked about any side effects you may have had.
* Blood (about 3 tablespoons) will be drawn for routine tests. If you are receiving everolimus, you will fast (have nothing to eat or drink except water) starting the night before these tests. The doctor will discuss this with you.
* Urine will be collected for routine tests if you are receiving everolimus or pazopanib.

Every 8 weeks, the following tests and procedures will be performed. If you are receiving the study treatment at your local doctor's office, you must return to MD Anderson for these tests and procedures.

* Blood (about 3 teaspoons) will be drawn for routine tests. If you are receiving pazopanib, this blood will also be used to check your thyroid function.
* You will have CT scans of the chest and abdomen to check the status of the disease.
* You will fill out 5 questionnaires about the quality of your life and about how you are feeling. This should take about 30 minutes.

Every year, you will have an MRI of the brain to check the status of the disease.

Every year, you will have an ECHO or MUGA scan to check the health of your heart.

Anytime the doctor decides it is needed, you will have scans such as a CT scan of the pelvis, an MRI scan of the abdomen or brain, ECHO or MUGA scan, and/or a bone scan.

After 1 year, if the disease has not gotten worse, you may have less clinic visits and tests.

Length of Participation:

You may continue taking a study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take a study drug if intolerable side effects occur, or if the disease gets worse after you take your second assigned study drug.

End-of-Treatment Visit:

When you are finished taking the study drug(s):

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking.
* You will be asked about any side effects you may have had.

Long-Term Follow-Up:

After your End-of-Treatment visit, the study staff will contact you by phone, e-mail, or you will come in for a clinic visit. You will be asked about how you are feeling and any side effects you may have had. Each follow-up will take about 5 minutes. Follow-up will take place every 3 months for the first 2 years, every 6 months for the third year, and 1 time a year after that. The last follow-up will be about 5 years after the last patient is enrolled.

This is an investigational study. Everolimus, bevacizumab, and pazopanib are all FDA approved and commercially available for kidney cancer. The investigational part of this study is to find out which order these drugs should be given in.

Up to 240 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed metastatic RCC with a clear cell component.
2. Prior radical or partial nephrectomy required. Patients whose primary tumor was treated with cryoablation or radiofrequency ablation would also be eligible.
3. Measurable disease
4. Age >/= 18 years. Because no dosing or adverse event data are currently available on the use of these targeted agents in patients < 18 years of age, children are excluded from this study
5. ECOG performance status 0 or 1
6. Adequate organ and marrow function within 14 days as defined below: a) Absolute neutrophil count /=> 1,500/microL; b) Platelets >/= 100,000/microL; c) Hgb >/= 9.0 g/dL (transfusion allowed); d) Total bilirubin < 1.5 mg/dl; e) Albumin > 2.5 g/dL; f) AST and ALT </= 2.5 X ULN for subjects without liver metastases; g) AST and ALT < 5 X ULN for subjects with liver metastases; h) Serum creatinine </= 2 mg/dL or CrCl >/= 50 cc/min; i) Fasting serum cholesterol </= 300 mg/dL or </= 7.75 mmol/L and fasting triglycerides </= 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
7. Female patients of childbearing potential must have a negative pregnancy test (serum/plasma or urine) within 7 days prior to beginning treatment on the study due to the possible teratogenic effect
8. Patients of child fathering or childbearing potential must agree to practice a form of medically acceptable birth control while on study
9. Patients must give written informed consent prior to initiation of study-related procedures. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy
10. Patients must be able to swallow pills
11. Both men and women and members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

1. No patient with any concurrent active malignancy, i.e. a patient requiring or receiving systemic therapy for another malignancy at the same time of treatment for RCC
2. Patients must not have received any prior targeted therapy (anti-VEGF agents or mTOR inhibitors), including adjuvant therapy, and must not have received any prior chemotherapy for mRCC. However, patients who had received prior immunotherapy, such as cytokines or vaccines, are permitted to enroll.
3. Patients must not be scheduled to receive another experimental drug while on this study. Patients are permitted to receive concomitant bisphosphonates.
4. Patients must not have multiple brain metastases or leptomeningeal disease. Patients with controlled solitary brain metastasis are eligible.
5. Patients must not have had a stroke or transient ischemic attack within 6 months.
6. Patients must not have uncontrolled infections.
7. Patients must not have clinically significant cardiovascular disease, defined as myocardial infarction (or unstable angina) within 6 months, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac dysrhythmia refractory to medical management
8. Patients must not have uncontrolled hypertension, defined as > 140/90 or prior history of hypertensive crisis or hypertensive encephalopathy. Treatment of hypertension with medications is permitted.
9. History of hemoptysis (>/= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
10. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
11. Symptomatic peripheral vascular disease
12. Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breast-feeding should be discontinued if the mother is enrolled on this trial.
13. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with some of these agents.
14. Patients must not have a clinical history of coagulopathy or bleeding diathesis. Patients may be on therapeutic anticoagulation preferably a low-molecular weight heparin. If the patients are on warfarin, the INR should be maintained within a therapeutic level and must be checked weekly for the first four weeks, then every 2 weeks for 4 additional weeks. Thereafter, they may be followed at the discretion of the treating provider. Antiplatelet agents are allowed.
15. Concomitant treatment with rifampin, St. John's wort, or the cytochrome p450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or Phenobarbital) is not allowed on this study.
16. Patients with significant baseline proteinuria defined as 300 or greater by screening U/A will be excluded if they have > 1,000 mg proteins in a 24-hour urine collection or if they have a random urine protein over creatinine (UPC) ratio >1.
17. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
18. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
19. Serious, non-healing wound, ulcer, or bone fracture
20. Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
21. Known hypersensitivity to any component of bevacizumab, pazopanib or everolimus.
22. Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
23. Patients with severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
24. Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C). Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
25. Patients receiving chronic, systemic treatment with steroids in pharmacological doses or immunosuppressive agents are excluded. Patients who receive steroids for physiological replacement, e.g., after adrenalectomy are not excluded. Topical or inhaled corticosteroids are also allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01-19 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to Overall Treatment Failure | 4 weeks
  Measured from date of randomization to date of second disease progression, 'drop-out' from protocol treatment for any reason or death, associated with each of the six two-agent sequential therapies given in parallel.

CONTACTS AND LOCATIONS:
Overall Officials: Amado Zurita, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org